CLINICAL TRIAL: NCT06095986
Title: A Proof of Concept, Prospective, Randomized, Placebo-controlled, Double-blind, Study to Evaluate the Safety, Tolerability, and Efficacy of Aramchol Meglumine in Patients With Primary Sclerosing Cholangitis
Brief Title: A Study Evaluating the Safety, Tolerability, and Efficacy of Aramchol Meglumine in Primary Sclerosing Cholangitis
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Operational and clinical reasons
Sponsor: Galmed Pharmaceuticals Ltd (Industry)
Collaborators: Virginia Commonwealth University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AM-002
Record Dates: First submitted 2023-10-11; First posted 2023-10-23 (Actual); Last update posted 2025-06-12 (Actual); Status verified 2025-06

CONDITIONS: Primary Sclerosing Cholangitis
MeSH Terms: conditions — Cholangitis, Sclerosing

STUDY DESIGN:
Intervention Model Description: Parallel group analysis
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double-blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- PSC patients administered with Aramchol meglumine (Active Comparator): Adult subjects with clinically diagnosed PSC that are administered with Aramchol meglumine
  Interventions: Drug: Aramchol meglumine
- PSC patients administered with placebo (Placebo Comparator): Adult subjects with clinically diagnosed PSC that are administered with matching placebo
  Interventions: Drug: Aramchol meglumine

INTERVENTIONS:
Drug: Aramchol meglumine — Aramchol meglumine is derived from a weak acid (Aramchol) and an amino-sugar (meglumine)

SUMMARY:
The objectives of this study is to Evaluate the Safety, Tolerability, and Efficacy of Aramchol Meglumine in Patients with Primary Sclerosing Cholangitis

DETAILED DESCRIPTION:
The objectives of this study are to:

* Establish the safety and tolerability of once daily (QD) Aramchol meglumine in patients with PSC
* Examine whether once daily (QD) Aramchol meglumine has any effect on serum alkaline phosphatase
* Provide a comprehensive readout of clinical efficacy following once daily (QD) Aramchol meglumine administration

ELIGIBILITY:
Inclusion Criteria:

1. Male or female age 18 years and above (inclusive at first screening visit)
2. Established diagnosis of large duct PSC based on abnormal cholangiography as assessed by magnetic resonance cholangiopancreatography (MRCP) or Endoscopic retrograde cholangiopancreatography (ERCP)
3. Alkaline phosphatase > 150 IU/l
4. Stable inflammatory bowel disease therapy > 3months for IBD patients
5. If receiving treatment with Ursodeoxycholic acid (UDCA; ursodiol), therapy is at a dose of <20 mg/kg/day, has been stable for at least 6 months before screening
6. Ability to understand the nature of the study and to sign a written informed consent form (ICF)

Exclusion Criteria:

1. Other causes of liver disease, including secondary sclerosing cholangitis or viral, metabolic, or alcoholic liver disease, as assessed clinically
2. Active Crohn's disease (CDAI > 40) or ulcerative colitis (Mayo IBD score > 4) or active non-hemorrhoidal rectal bleeding
3. Small bowel resection > 100 cm
4. Cirrhosis (clinically evident or by biopsy)
5. Prior hepatic decompensation event
6. Recent (< 6 weeks) acute cholangitis or hospitalization for PSC or IBD
7. Bleeding diathesis or other contraindication for liver biopsy
8. Known GI or hepatobiliary malignancy
9. Prior liver transplantation
10. Prior exposure to study drug
11. Active untreated viral hepatitis or other concomitant liver disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2025-06 (Estimated); Primary Completion 2026-09 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline in serum alkaline phosphatase (ALP) | 48 weeks
  The change from Baseline to Week 48 in ALP levels

SECONDARY OUTCOMES:
Change from Baseline in hepatobiliary fibrosis using the Nakanuma staging scale | 48 weeks
  Change from Baseline to Week 48 in liver histology using the Nakanuma stage classification. A score of 0 is classified as stage 1 (no or minimal disease progression), while 1 score 5 or 6 is classified as stage 4 (advanced disease progression).
Change from Baseline in Enhanced liver fibrosis (ELF) | 48 weeks
  Change from Baseline to Week 48 in Enhanced liver fibrosis (ELF) test. Score below 7.7 indicate no to mild fibrosis, and score higher than 11.3 indicate cirrhosis.
Change from Baseline in MRCP | 48 weeks
  Change from Baseline to Week 48 in magnetic resonance cholangiopancreatography (MRCP)
Change from Baseline in quantitative liver function using Gadoxetate clearance | 48 weeks
  Change from Baseline to Week 48 in quantitative liver function using Gadoxetate clearance
Change from Baseline in 5D-itch scale | 48 weeks
  Change from Baseline to Week 48 in the 5 dimension itch scale (5d-itch scale) measuring pruritus (the 5 dimensions are degree, duration, direction, disability and distribution). Higher degree mean worse outcome <8 on rating scale mean no pruritus, and >22 on rating scale indicate severe pruritus
Change from Baseline to Week 48 in Patient-Reported Outcomes Measurement Information System (PROMIS)-19 score | 48 weeks
  Change from Baseline to Week 48 in the Patient-Reported Outcomes Measurement Information System (PROMIS)-19 questionnaire score. The average score for Physical Function is 50, with a score of 40 considered below average and a score of 60 considered above average
Change from Baseline in the Mayo IBD symptom severity score | 48 weeks
  Change from Baseline to Week 48 in the Mayo Inflammatory bowel disease (IBD) symptom severity score. A score of 3 to 5 points indicates mildly active disease and a score of 11 to 12 points indicates severely active bowel disease
Change from Baseline in the revised Mayo risk score (rMRS) | 48 weeks
  Change from Baseline to Week 48 in the revised Mayo risk score (rMRS). The score provide the estimated probability of survival (%) based on age, bilirubin, AST, and history of bleeding
Change from Baseline in the UK-PSC score | 48 weeks
  Change from Baseline to Week 48 in the united kingdom primary sclerosing cholangitis (UK-PSC) score. The score provide the estimated probability of survival (%) based on age, bilirubin, albumin, platelets, hemoglobin and ALP
Change from Baseline in the PSC risk estimate tool (PREsTo) | 48 weeks
  Change from Baseline to Week 48 in the PSC risk estimate tool (PREsTo). The tool consists of bilirubin, albumin, ALP, platelets, AST, hemoglobin, sodium, patient age and the number of years since PSC was diagnosed, and it predicts short-term and long-term need for liver transplantation or death.

CONTACTS AND LOCATIONS:
Overall Officials: Arun Sanyal, MD, Principal Investigator — The Sanyal Institute for Liver Disease & Metabolic Health at VCU
Locations (1):
- The Sanyal Institute for Liver Disease & Metabolic Health at VCU, Richmond, Virginia, United States

IPD SHARING:
Plan to Share IPD: Yes
Share the study protocol and SAP
Supporting Information: Study Protocol, SAP
Time Frame: Study completion
Access Criteria: Any person with access to ClinicalTrials.gov
URL: https://galmedpharma.com/